CLINICAL TRIAL: NCT00037310
Title: New CVD Risk Factors for Lowered Cognitive Functioning
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1161; R01HL067358 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Neurologic Manifestations
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Neurologic Manifestations

SUMMARY:
To explore the associations between cognitive functioning and three major cardiovascular disease risk factors: high blood pressure; high total plasma homocysteine (tHcy); and ApoE e4 genotype.

DETAILED DESCRIPTION:
BACKGROUND:

Arterial hypertension and high blood pressure (HBP) are major risk factors for cardiovascular disease (CVD) and stroke; they are also risk factors for lowered cognitive functioning. Except for diabetes, there have been comparatively few studies of other common risk factors, particularly with regard to interrelationships among risk factors which may adversely affect cognitive ability.

DESIGN NARRATIVE:

The study examines associations between cognitive functioning and three cardiovascular risk factors: 1) high blood pressure; 2) high total plasma homocysteine (tHcy), and 3) ApoE e4 genotype. These associations are examined cross-sectionally as well as longitudinally, using data collected at a follow-up visit of members of a cohort that has been followed for the past 18-19 years. Longitudinal data are used to examine both current and change in cognitive functioning. Some analyses are prospective (e.g., high blood pressure and change in cognitive functioning), while others are cross-sectional (e.g., ApoE e4 and current cognitive functioning) or retrospective (e.g., tHcy and change in cognitive functioning). Structural equation models are used to examine cross-sectional data in elucidating a general theoretical model. Two-stage growth curve analyses and survival analyses are appropriate methods for analyzing the longitudinal data. The study includes a very comprehensive set of measures that have already been collected or will be collected during the follow-up visit. All potential confounders of the association between the three target predictor variables and the various domains of cognitive functioning appear to have been included in this design.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merrill Elias — University of Maine

REFERENCES:
- [Background] Elias PK, Elias MF, Robbins MA, Budge MM. Blood pressure-related cognitive decline: does age make a difference? Hypertension. 2004 Nov;44(5):631-6. doi: 10.1161/01.HYP.0000145858.07252.99. Epub 2004 Oct 4. PMID 15466661